CLINICAL TRIAL: NCT04511468
Title: A Combination of Zinc, Chromium, Vitamin C, and Copper Supplement for Prediabetes Progression: Randomized Controlled-Trial in Jakarta
Brief Title: Zinc, Chromium, Vitamin C, and Copper Combination Supplement for Prediabetes Progression
Acronym: CHANGE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Blackmores Institute (Industry)
Responsible Party: Principal Investigator, Prof Rina Agustina, MD, PhD, dr. Rina Agustina, M.Sc., PhD, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CHANGE
Record Dates: First submitted 2020-06-01; First posted 2020-08-13 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: PreDiabetes; Nutrition
Keywords: Zinc; Chromium; Copper; Vitamin C
MeSH Terms: conditions — Prediabetic State | interventions — Zinc; Chromium; Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: There will be two arms of intervention:
  Arm 1: A combination of Zinc, Chromium, Vitamin C, and Copper (ZCC supplement) with standard healthy lifestyle intervention.
  Arm 2: A combination of placebo with standard healthy lifestyle intervention.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Independent party will mask the product.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): A combination of Zinc, Chromium, Vitamin C, and Copper (ZCC supplement) with standard healthy lifestyle intervention
  Interventions: Dietary Supplement: Zinc, Chromium, Vitamin C, and Copper Supplementation; Behavioral: Standard healthy lifestyle intervention
- Control group (Placebo Comparator): Placebo with standard healthy lifestyle intervention
  Interventions: Behavioral: Standard healthy lifestyle intervention; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Zinc, Chromium, Vitamin C, and Copper Supplementation — Combination of mineral and vitamin supplementation that consist of Zinc, Chromium, Vitamin C, and Copper
  Arms: Experimental Group
Behavioral: Standard healthy lifestyle intervention — Standard healthy lifestyle intervention will follow the Guidelines on the Management and Prevention of Prediabetes by the Indonesian Ministry of Healthy and the Indonesian Diabetes Association.
Other: Placebo — Placebo with inactive ingredients
  Arms: Control group

SUMMARY:
Currently, the incidence of diabetes mellitus is increasing worldwide. People with prediabetes have higher risk to develop diabetes mellitus type 2. Several studies have proven that Zinc and Chromium are minerals that contribute to decreasing the level of blood glucose and insulin resistance. In addition, vitamin C also contributes in decreasing Fasting Blood Glucose (FBG) and Hemoglobin A1c (HbA1c). However, the eficacy of a combined zinc, chromium, vitamin C, and copper (ZCC) in decreasing blood glucose in prediabetic people has never been performed.

The primary objective of this study is to investigate the effect of a combination of ZCC supplementation with standard healthy lifestyle counseling in improving glucose profile [Fasting Blood Glucose (FBG), 2-hour Oral Glucose Tolerance Test (OGTT), Homeostatic Model Assessment for Insulin Resistance (HOMA-IR)] from prediabetes to normal or reducing the risk of progression from prediabetes to Type 2-Diabetes Mellitus (T2DM) compared to placebo with standard healthy lifestyle intervention.

DETAILED DESCRIPTION:
Diabetes is an important public health problem as the number of people with diabetes are increasing across the world and contributes to high mortality burden. Prediabetes is an intermediate stage between normal glucose tolerance and type 2 diabetes mellitus. Furthermore, people with prediabetes have higher risk to develop diabetes mellitus type 2.

There are several objectives in this study, such as primary objective, secondary objectives, and exploratory objectives.

1. Primary Objective:

   To investigate the effect of a combination of Zinc, Chromium, Vitamin C, and Copper supplementation (ZCC supplementation) with standard healthy lifestyle intervention in improving glucose profile [Fasting Blood Glucose (FBG), 2-hour Oral Glucose Tolerance Test (OGTT), Homeostatic Model Assessment for Insulin Resistance (HOMA-IR)]) from prediabetes to normal (reducing the proportion of prediabetes and increasing the proportion to become normal) or reducing the risk of progression from prediabetes to Type 2-Diabetes Mellitus (T2DM) compared to placebo with standard healthy lifestyle intervention.
2. Secondary Objectives:

   To investigate the level of Zinc and Chromium among the prediabetes, the safety of the ZCC supplementation, and the effect of a combination of Zinc, Chromium, Vitamin C, and Copper supplementation (ZCC supplementation) among prediabetic adults compared to the placebo supplementation on:
   1. Lipid profile [Low-Density Lipoprotein (LDL), High-Density Lipoprotein (HDL), Triglyceride];
   2. Hemoglobin A1c (HbA1c);
   3. Dietary intake and physical activity
   4. Body weight and composition (body weight, Body Mass Index (BMI), body fat).
3. Exploratory Objectives:

   1. To determine cost effectiveness of intervention on prediabetic adults comparing two different intervention models
   2. To determine the quality of life of prediabetes adults receiving a combination of zinc, chromium, vitamin C, and copper supplementation.
   3. Level of hs-crp; TNF-alpha and Vitamin C will be assessed later if needed (optional)

Study Design:

This study is a double-blind, randomized, placebo-controlled trial in the community setting, with two arms of intervention involving a total of 670 people.

Study Duration:

This study is a two-year study with 1 year of intervention for each subject.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 35-65 years old;
* Being prediabetes as assessed by having fasting plasma glucose (FPG) level in the range of 100 mg/dL to 125 mg/dL; having 2-h values in the oral glucose tolerance (OGTT) level in the range of 140 mg/dL to 199 mg/dL;
* The study subjects will be recruited from household communities connected to any health care facilities such as primary health center, private clinics or private GP/specialist on the national health care system;
* The subjects are willing to sign informed consent;
* The subjects are willing to stay commitment during the study, at least 1 year;
* Having app-android mobile

Exclusion Criteria:

* Pregnancy or lactation women;
* Transgender on hormonal injection;
* Bariatric surgery;
* Consuming other pills supplementation containing zinc and/or chromium, copper, vitamin C in regular basis;
* History of Inflammatory Bowel Disease (IBD), psychiatric disorders, chronic diseases (e.g., HIV, Cushing syndrome, CKD, acromegaly, hyperthyroidism, etc.);
* Not healthy (current status of the severely malnourished, acute problem of any severe disease, history of impaired hepatic, renal failure, heart failure, cancer, other catastrophic diseases.
* Currently using weight loss medication;
* Consuming pharmacology agents that might interfere the intervention (such as metformin, methylprednisolone, methyltestosterone, diuretics, complementary medicines);
* Subjects who are unable to read and understand the statements of consent form

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 670 (Estimated)
Dates: Start 2021-06-23 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change of Fasting Blood Glucose (FBG) | Baseline (at the beginning of study), Intervention Period (3 and 6 months), and 12 months
  To investigate the effect of ZCC supplementation with standard healthy lifestyle intervention in improving Fasting Blood Glucose compared to placebo with standard healthy lifestyle intervention
Change of Hemoglobin A1c (HbA1c) | Baseline (at the beginning of study), Intervention Period (3 and 6 months), and 12 months
  To investigate the effect of ZCC supplementation with standard healthy lifestyle intervention in improving HbA1c compared to placebo with standard healthy lifestyle intervention
Change of 2 hour Oral Glucose Tolerance Test (2-hour OGTT) | Baseline (at the beginning of study), Intervention Period (3 and 6 months), and 12 months
  To investigate the effect of ZCC supplementation with standard healthy lifestyle intervention in improving 2 hour OGTT compared to placebo with standard healthy lifestyle intervention
Change of Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | Baseline (at the beginning of study), Intervention Period (3 and 6 months), and 12 months
  To investigate the effect of ZCC supplementation with standard healthy lifestyle intervention in improving HOMA-IR compared to placebo with standard healthy lifestyle intervention
Delay Onset of Type 2 Diabetes Mellitus (T2DM) Progression | Baseline (at the beginning of study), Intervention Period (3 and 6 months), and 12 months
  Total participants who develop T2DM during study intervention as assessed by blood glucose
Change the Risk of T2DM Progression | Baseline (at the beginning of study), Intervention Period (3 and 6 months), and 12 months
  Total participants whose blood glucose returned to normal during study intervention as assessed by blood glucose

SECONDARY OUTCOMES:
Change in Lipid Profile (will be assessed by High Density Lipoprotein (HDL) in mg/dL, Low Density Lipoprotein (LDL) in mg/dL, Triglyceride (TG) in mg/dL, and total cholesterol in mg/dL)) | Baseline (at the beginning of study), Intervention Period (3 and 6 months), and 12 months
  To investigate the effect of ZCC supplementation among prediabetes adults on lipid profile (HDL, LDL, TG and total cholesterol)
Change in Body Weight (kilogram) | Baseline (at the beginning of study), Intervention Period (3 and 6 months), and 12 months
  To investigate the effect of ZCC supplementation among prediabetes adults on changing in body weight.
Change in Body Mass Index (BMI) (weight and height will be combined to report the BMI in kg/m^2) | Baseline (at the beginning of study), Intervention Period (3 and 6 months), and 12 months
  To investigate the effect of ZCC supplementation among prediabetes adults on changing in BMI.
Change in Percentage of Fat Mass (using Body Impedance Analysis) | Baseline (at the beginning of study), Intervention Period (3 and 6 months), and 12 months
  To investigate the effect of ZCC supplementation among prediabetes adults on changing in fat mass using Body Impedance Analysis.
Change in Dietary intake | Baseline (at the beginning of study), Intervention Period (3 and 6 months), and 12 months
  To determine the differences in changes of dietary intake after receiving 12 months of ZCC or placebo supplementation with standard healthy lifestyle intervention.
The Difference of Zinc Level among prediabetes adults | Baseline (at the beginning of study)
  To determine the difference of Zinc level in prediabetes adults.
The Difference of Chromium Level among prediabetes adults | Baseline (at the beginning of study)
  To determine the difference of Chromium level in prediabetes adults.
Change in Physical Activity (assessed by IPAQ Questionnaire) | Baseline (at the beginning of study), Intervention Period (3 and 6 months), and 12 months
  To determine the difference of physical activity in prediabetes adults using standardized questionnaire on control and intervention group. Moderate intensity activities have been established as between 3 and 6 METS (metabolic equivalent of task). One MET is the amount of energy used while sitting quietly. Physical activities will be rated using METs to indicate their intensity. Vigorous-intensity activity activities have been established as >6 METs. The higher the MET scores mean a better physical activity.
The assessment on the Safety of the ZCC Supplementation for the respondents | Baseline (at the beginning of study) and 12 months (end of the study)
  To investigate the safety of the ZCC supplementation among prediabetes adults on the kidney function, liver function, and complete peripheral blood to assess whether the supplements have the specific effects for the respondents' organ function.

OTHER OUTCOMES:
Cost Effectiveness Analysis of ZCC Supplement using Incremental cost-effectiveness ratio (ICER) | through study completion, an average of 1 year
  Analyzing the cost effectiveness of intervention on Prediabetic adults comparing 2 different intervention models using incremental cost-effectiveness ratio (ICER). ICER is the ratio of the change in costs of a therapeutic intervention (compared to the alternative, such as doing nothing or using the best available alternative treatment) to the change in effects of the intervention.
Change of Quality of Life Questionnaire (assessed by SF-36 questionnaire) | through study completion, an average of 1 year
  To determine the quality of life of prediabetes adults using standardized questionnaire on control and intervention group. he range of scores is between 15 to 105, with a higher score or number being indicative of a higher quality of life.
Change in High-sensitivity C-Reactive Protein (hs-CRP) level (optional) | through study completion, an average of 2 year
  To determine the difference of hs-CRP level in prediabetes adults with ZCC and placebo supplementation (optional).
Change in Tumor Necrosis Factor-alpha (TNF-alpha) Level (optional) | through study completion, an average of 2 year
  To determine the difference of TNF-alpha level in prediabetes adults with ZCC and placebo supplementation (optional).
Change in Vitamin C Level (optional) | through study completion, an average of 2 year
  To determine the difference of Vitamin C level in prediabetes adults with ZCC and placebo supplementation (optional).

CONTACTS AND LOCATIONS:
Overall Officials: Rina Agustina, MD, MSc, PhD, Principal Investigator — HNRC-IMERI, Faculty of Medicine Universitas Indonesia
Locations (1):
- Human Nutrition Research Center, Indonesian Medical Education Research Institute (HNRC-IMERI) Faculty of Medicine, Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jayawardena R, Ranasinghe P, Byrne NM, Soares MJ, Katulanda P, Hills AP. Prevalence and trends of the diabetes epidemic in South Asia: a systematic review and meta-analysis. BMC Public Health. 2012 May 25;12:380. doi: 10.1186/1471-2458-12-380. PMID 22630043
- [Background] Jayawardena R, Ranasinghe P, Galappatthy P, Malkanthi R, Constantine G, Katulanda P. Effects of zinc supplementation on diabetes mellitus: a systematic review and meta-analysis. Diabetol Metab Syndr. 2012 Apr 19;4(1):13. doi: 10.1186/1758-5996-4-13. PMID 22515411
- [Background] Dall TM, Yang W, Gillespie K, Mocarski M, Byrne E, Cintina I, Beronja K, Semilla AP, Iacobucci W, Hogan PF. The Economic Burden of Elevated Blood Glucose Levels in 2017: Diagnosed and Undiagnosed Diabetes, Gestational Diabetes Mellitus, and Prediabetes. Diabetes Care. 2019 Sep;42(9):1661-1668. doi: 10.2337/dc18-1226. Epub 2019 Apr 2. PMID 30940641
- [Background] Janghorbani M, Amini M. Normal fasting plasma glucose and risk of prediabetes and type 2 diabetes: the Isfahan Diabetes Prevention Study. Rev Diabet Stud. 2011 Winter;8(4):490-8. doi: 10.1900/RDS.2011.8.490. Epub 2012 Feb 10. PMID 22580730
- [Background] Aroda VR, Ratner R. Approach to the patient with prediabetes. J Clin Endocrinol Metab. 2008 Sep;93(9):3259-65. doi: 10.1210/jc.2008-1091. PMID 18772457
- [Background] Kelly FJ. Use of antioxidants in the prevention and treatment of disease. J Int Fed Clin Chem. 1998 Mar;10(1):21-3. PMID 10181011
- [Background] Capdor J, Foster M, Petocz P, Samman S. Zinc and glycemic control: a meta-analysis of randomised placebo controlled supplementation trials in humans. J Trace Elem Med Biol. 2013 Apr;27(2):137-42. doi: 10.1016/j.jtemb.2012.08.001. Epub 2012 Nov 6. PMID 23137858
- [Background] Ranasinghe P, Wathurapatha WS, Galappatthy P, Katulanda P, Jayawardena R, Constantine GR. Zinc supplementation in prediabetes: A randomized double-blind placebo-controlled clinical trial. J Diabetes. 2018 May;10(5):386-397. doi: 10.1111/1753-0407.12621. Epub 2018 Jan 3. PMID 29072815
- [Background] Guo CH, Wang CL. Effects of zinc supplementation on plasma copper/zinc ratios, oxidative stress, and immunological status in hemodialysis patients. Int J Med Sci. 2013;10(1):79-89. doi: 10.7150/ijms.5291. Epub 2012 Dec 22. PMID 23289009
- [Background] Kim HN, Kim SH, Eun YM, Song SW. Effects of zinc, magnesium, and chromium supplementation on cardiometabolic risk in adults with metabolic syndrome: A double-blind, placebo-controlled randomised trial. J Trace Elem Med Biol. 2018 Jul;48:166-171. doi: 10.1016/j.jtemb.2018.03.022. Epub 2018 Mar 30. PMID 29773176
- [Background] Bartlett HE, Eperjesi F. Nutritional supplementation for type 2 diabetes: a systematic review. Ophthalmic Physiol Opt. 2008 Nov;28(6):503-23. doi: 10.1111/j.1475-1313.2008.00595.x. PMID 19076553
- [Background] Abdollahi M, Farshchi A, Nikfar S, Seyedifar M. Effect of chromium on glucose and lipid profiles in patients with type 2 diabetes; a meta-analysis review of randomized trials. J Pharm Pharm Sci. 2013;16(1):99-114. doi: 10.18433/j3g022. PMID 23683609
- [Background] Will JC, Ford ES, Bowman BA. Serum vitamin C concentrations and diabetes: findings from the Third National Health and Nutrition Examination Survey, 1988-1994. Am J Clin Nutr. 1999 Jul;70(1):49-52. doi: 10.1093/ajcn/70.1.49. PMID 10393138
- [Background] Eriksson J, Kohvakka A. Magnesium and ascorbic acid supplementation in diabetes mellitus. Ann Nutr Metab. 1995;39(4):217-23. doi: 10.1159/000177865. PMID 8546437
- [Background] Ashor AW, Werner AD, Lara J, Willis ND, Mathers JC, Siervo M. Effects of vitamin C supplementation on glycaemic control: a systematic review and meta-analysis of randomised controlled trials. Eur J Clin Nutr. 2017 Dec;71(12):1371-1380. doi: 10.1038/ejcn.2017.24. Epub 2017 Mar 15. PMID 28294172
- [Background] Islam MR, Attia J, Ali L, McEvoy M, Selim S, Sibbritt D, Akhter A, Akter S, Peel R, Faruque O, Mona T, Lona H, Milton AH. Zinc supplementation for improving glucose handling in pre-diabetes: A double blind randomized placebo controlled pilot study. Diabetes Res Clin Pract. 2016 May;115:39-46. doi: 10.1016/j.diabres.2016.03.010. Epub 2016 Mar 19. PMID 27242121
- [Background] Sharma S, Agrawal RP, Choudhary M, Jain S, Goyal S, Agarwal V. Beneficial effect of chromium supplementation on glucose, HbA1C and lipid variables in individuals with newly onset type-2 diabetes. J Trace Elem Med Biol. 2011 Jul;25(3):149-53. doi: 10.1016/j.jtemb.2011.03.003. Epub 2011 May 12. PMID 21570271
- [Background] Paiva AN, Lima JG, Medeiros AC, Figueiredo HA, Andrade RL, Ururahy MA, Rezende AA, Brandao-Neto J, Almeida Md. Beneficial effects of oral chromium picolinate supplementation on glycemic control in patients with type 2 diabetes: A randomized clinical study. J Trace Elem Med Biol. 2015 Oct;32:66-72. doi: 10.1016/j.jtemb.2015.05.006. Epub 2015 May 28. PMID 26302914
- [Background] Vistisen D, Kivimaki M, Perreault L, Hulman A, Witte DR, Brunner EJ, Tabak A, Jorgensen ME, Faerch K. Reversion from prediabetes to normoglycaemia and risk of cardiovascular disease and mortality: the Whitehall II cohort study. Diabetologia. 2019 Aug;62(8):1385-1390. doi: 10.1007/s00125-019-4895-0. Epub 2019 May 23. PMID 31123789
- [Background] Khan MI, Siddique KU, Ashfaq F, Ali W, Reddy HD, Mishra A. Effect of high-dose zinc supplementation with oral hypoglycemic agents on glycemic control and inflammation in type-2 diabetic nephropathy patients. J Nat Sci Biol Med. 2013 Jul;4(2):336-40. doi: 10.4103/0976-9668.117002. PMID 24082728
- [Derived] Agustina R, Prafiantini E, Putri AR, Mufida R, Hanifa H, Afifah S, Tahapary DL, Shankar AH, Soewondo P. Protocol for a randomized controlled trial to evaluate the impact of daily supplementation with zinc, chromium, vitamin C, and copper on progression of prediabetes in Jakarta, Indonesia. Contemp Clin Trials. 2025 Sep;156:108007. doi: 10.1016/j.cct.2025.108007. Epub 2025 Jul 11. PMID 40653308